CLINICAL TRIAL: NCT00414700
Title: Prospective Multicenter Randomized Controlled Trial of ChondroCelect® (Via Autologous Chondrocyte Implantation) vs Microfracture (as Procedure) in the Repair of Symptomatic Cartilaginous Defects of the Femoral Condyles
Brief Title: RCT of ChondroCelect® (in an ACI Procedure) vs Microfracture in the Repair of Cartilage Defects of the Knee
Acronym: TIGACT01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TiGenix n.v. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TIG/ACT/01/2000&Extension; BB IND 12491 0007 (Other: CBER)
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Articular Cartilage Lesion of the Femoral Condyle
Keywords: Cartilage; Articular; Femoral; Knee
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ChondroCelect (Experimental)
  Interventions: Drug: ChondroCelect implantation
- Microfracture (Active Comparator)
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Drug: ChondroCelect implantation — 10.000 cells/µl cell suspension for implantation (Autologous Chondrocyte Implantation). ChondroCelect consists of characterised autologous cartilage-forming cells expressing a specific marker profile.
  The dose depends on the size of the lesion. Recommended dose is 0.8 to 1.0 million cells/cm².
  Other Names: CCI
  Arms: ChondroCelect
Procedure: Microfracture — A procedure in which the subchondral bone is perforated to allow a bloodcloth to form scar tissue.
  Other Names: subchondral drilling
  Arms: Microfracture

SUMMARY:
This is a phase III, multicenter, open-label, randomized controlled trial of ChondroCelect® in an Autologous Chondrocyte Implantation (ACI) procedure compared to the procedure of microfracture (MF) in the repair of symptomatic cartilage lesions of the knee. Eligible patients attended two screening visits and were booked for arthroscopy approximately 2 weeks later. At that time, patients were randomized to either ACI with ChondroCelect® or to MF, a procedure in which the subchondral bone is perforated to allow a bloodcloth to form scar tissue. Patients randomized to MF had the procedure performed at the time of their arthroscopy; those randomized to ACI with ChondroCelect® had their cells harvested during the arthroscopy and then returned to the clinic approximately 4 weeks later for an open knee procedure, during which the ACI procedure using ChondroCelect® was performed. Patients subsequently followed the same rehabilitation program and had follow-up assessments up to 12 months post-surgery. The 12-month visit was the end-of-study visit for the TIG/ACT/01/2000 protocol. Subject to satisfying the eligibility criteria, patients who had participated in the initial 12 month trial could enter the extension trial. The 12-month visit for the initial study was the baseline visit for the extension study. During the extension study, patients have follow-up assessments up to 60 months post-surgery.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* Signed patient informed consent
* Symptomatic cartilage single lesion of the femoral condyle
* Lesion on femoral condyle between 1 and 5 cm²
* Agree to participate actively in a strict rehabilitation protocol and follow-up programme
* Agree to only use paracetamol mono-or combination preparation (max 4g/d) and Non-Steroidal Anti Inflammatory Drugs (NSAIDS) during the study and to discontinue this medication 2 weeks before the baseline visit and the follow-up visits. The use of paracetamol mono-preparation (max 4g/d) is allowed up to one week before the baseline visit and the follow-up visits.
* Females of childbearing age should use a proven method to prevent pregnancy

Exclusion Criteria:

* Participation in concurrent trials
* Participation in previous trials within 3 months
* Subjects with hepatitis, HIV or syphilis
* Malignancy
* Alcohol or drug (medication) abuse
* Poor general health as judged by Investigator
* Clinically relevant second cartilage lesion on the patella
* Patellofemoral cartilage lesion
* Osteochondritis Dissecans (OCD) : recent OCD (within 1 year before baseline), depth of lesion > 0.5cm, subchondral slerosis
* Advanced osteoarthritis (OA) : radiographic atlas of OA grade 2-3
* Known allergy to gentamicin or penicillins (or presence of multiple severe allergies)
* Complex ligamentous instability of the knee
* Meniscal transplant
* Meniscal suture with meniscal arrows (ipsilateral)
* Meniscus resection : if < 1 yr before baseline - lateral meniscus resection or medial meniscus resection of more than 50%. If > 1 yr before baseline - ipsilateral meniscus resection of more than 50%, controlateral meniscus resection of more than 50% if ipsilateral meniscus is not intact, combination of medial and lateral meniscus resection and one of both > 50%.
* Varus or valgus malalignment of more than 5°
* Mosaicplasty
* Microfracture performed less than 1 yr before baseline
* Having received hyaluronic acid intra-articular injections in the affected knee within the last 6 months of baseline
* Taking specific OA drugs such as chondroïtin sulfate, diacerein, n-glucosamine, piascledine, capsaicin within 2 weeks of the baseline visit
* Corticosteroïd treatment by systemic or intra-articular route within the last month of baseline or intramuscular or oral corticosteroïds within the last 2 weeks of baseline
* Chronic use of anticoagulants
* Uncontrolled diabetes
* Any concomitant painful or disabling disease of the spine,hips or lower limbs that would interfere with evaluation of the afflicted knee
* Any clinically significant or symptomatic vascular or neurologic disorder of the lower extremities
* Any evidence of the following diseases in the target joint : septic arthritis, inflammatory joint disease, gout, recurrent episodes of pseudogout, Paget's disease of bone, ochronosis, acromegaly, hemochromatosis, Wilson's disease, primary osteochondromatosis, heritable disorders, collagen gene mutation
* Current diagnosis of osteomyelitis
* Liver enzymes (SGOT, SGPT, Alkaline Phosphatase) of more then two times the upper limit of normal or any other result that is clinically important according to the Investigator
* CRP > 10 mg/l

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2002-02; Primary Completion 2006-07 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniël BF Saris, M.D., Ph.D., Principal Investigator — University Medical Center Utrecht, Department of Orthopedics, Heidelberglaan 100, 3584 CX Utrecht, The Netherlands.; Johan Vanlauwe, M.D., Principal Investigator — University Hospitals Leuven, Department of Orthopedics, Herestraat 49, 3000 Leuven, Weligerveld 1, 3212 Pellenberg, Belgium.; Frank P Luyten, M.D., Ph.D., Study Director — Division of Rheumatology, Department of Muskuloskeletal Sciences, University Hospitals, Katholieke Universiteit Leuven, Herestraat 49, 3000 Leuven, Belgium
Locations (12):
- Belgium (9):
  - AZ St. Jan Brugge, Department of Orthopedics, Bruges
  - AZ St Lucas Brugge, Department of Orthopedics, Bruges
  - Academisch Ziekenhuis, Vrije Universiteit Brussel, Department of Orthopedics, Brussels
  - SPM Monica Antwerp, Deurne
  - Ghent University Hospital, Department of Orthopedics, Ghent
  - AZ St. Elisabeth, Department of Orthopedics, Herentals
  - AZ Groeninge, Department of Orthopedics, Kortrijk
  - University Hospitals Leuven, Department of Orthopedics, Leuven
  - A.Z. Sint Jozef, Department of Orthopedics, Malle
- Department of Orthopedic Surgery, School of Medicine, University of Zagreb, Zagreb, Croatia
- University Hospital Hannover, Department of Orthopedics, Hanover, Germany
- University Medical Center Utrecht, Department of Orthopedics, Utrecht, Netherlands

REFERENCES:
- [Background] Dell'Accio F, Vanlauwe J, Bellemans J, Neys J, De Bari C, Luyten FP. Expanded phenotypically stable chondrocytes persist in the repair tissue and contribute to cartilage matrix formation and structural integration in a goat model of autologous chondrocyte implantation. J Orthop Res. 2003 Jan;21(1):123-31. doi: 10.1016/S0736-0266(02)00090-6. PMID 12507589
- [Background] Dell'Accio F, De Bari C, Luyten FP. Microenvironment and phenotypic stability specify tissue formation by human articular cartilage-derived cells in vivo. Exp Cell Res. 2003 Jul 1;287(1):16-27. doi: 10.1016/s0014-4827(03)00036-3. PMID 12799178
- [Background] Dell'Accio F, De Bari C, Luyten FP. Molecular markers predictive of the capacity of expanded human articular chondrocytes to form stable cartilage in vivo. Arthritis Rheum. 2001 Jul;44(7):1608-19. doi: 10.1002/1529-0131(200107)44:73.0.CO;2-T. PMID 11465712
- [Background] Brittberg M, Lindahl A, Nilsson A, Ohlsson C, Isaksson O, Peterson L. Treatment of deep cartilage defects in the knee with autologous chondrocyte transplantation. N Engl J Med. 1994 Oct 6;331(14):889-95. doi: 10.1056/NEJM199410063311401. PMID 8078550
- [Background] Knutsen G, Engebretsen L, Ludvigsen TC, Drogset JO, Grontvedt T, Solheim E, Strand T, Roberts S, Isaksen V, Johansen O. Autologous chondrocyte implantation compared with microfracture in the knee. A randomized trial. J Bone Joint Surg Am. 2004 Mar;86(3):455-64. doi: 10.2106/00004623-200403000-00001. PMID 14996869
- [Background] Rosenzweig A. Cardiac cell therapy--mixed results from mixed cells. N Engl J Med. 2006 Sep 21;355(12):1274-7. doi: 10.1056/NEJMe068172. No abstract available. PMID 16990391
- [Result] Saris DB, Vanlauwe J, Victor J, Haspl M, Bohnsack M, Fortems Y, Vandekerckhove B, Almqvist KF, Claes T, Handelberg F, Lagae K, van der Bauwhede J, Vandenneucker H, Yang KG, Jelic M, Verdonk R, Veulemans N, Bellemans J, Luyten FP. Characterized chondrocyte implantation results in better structural repair when treating symptomatic cartilage defects of the knee in a randomized controlled trial versus microfracture. Am J Sports Med. 2008 Feb;36(2):235-46. doi: 10.1177/0363546507311095. PMID 18202295
- [Result] Saris DB, Vanlauwe J, Victor J, Almqvist KF, Verdonk R, Bellemans J, Luyten FP; TIG/ACT/01/2000&EXT Study Group. Treatment of symptomatic cartilage defects of the knee: characterized chondrocyte implantation results in better clinical outcome at 36 months in a randomized trial compared to microfracture. Am J Sports Med. 2009 Nov;37 Suppl 1:10S-19S. doi: 10.1177/0363546509350694. Epub 2009 Oct 21. PMID 19846694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment by orthopaedic surgeons (medical clinic). Recruitment period: 21 February 2002 to 23 November 2004.
Pre-assignment Details: Enrolled patients excluded: Not fulfilling inclusion criteria. Withdrawal of consent.
Groups:
- ChondroCelect: ChondroCelect is intended for use in autologous cartilage repair and is administered to patients in an Autologous Chondrocyte Implantation procedure (ACI)
- Microfracture: Microfracture is a surgical technique involving several systematic steps, including debridement to a stable cartilage margin, careful removal of the calcified cartilage layer, and homogeneous placement of microfracture penetrations within the cartilage defect with resultant complete defect fill by a well-anchored mesenchymal clot.
Period: Overall Study
Arm/Group | ChondroCelect | Microfracture
Started | 57 | 61
Completed | 51 | 58
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ChondroCelect | Microfracture | Total
Number analyzed (Participants) | 57 | 61 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 61 | 118
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33.93 (8.54) | 33.92 (8.61) | 33.92 (8.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 35 | 41 | 76
Region of Enrollment [Number; unit: participants]
  Belgium | 33 | 35 | 68
  Croatia | 4 | 5 | 9
  Germany | 1 | 4 | 5
  Netherlands | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Histomorphometry Safranin-O + Anti-Collagen II Antibody Staining
Description: Histomorphometry on end point biopsies at 12 months post-surgery. Safranin-O (ratio 0-1)+ anti-Collagen II antibody (ratio 0-1) stain signal expressed as a ratio of the total cartilage surface area (Saf O + anti Coll II divided by total surface = ratio 0-2). Safranin-O stains proteoglycans and anti-Collagen II antibody reflects the presence of Collagen II.
Time Frame: 12 months post-surgery
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | ChondroCelect | Microfracture
Number analyzed (Participants) | 51 | 58
Ratio | 1.01 (0.08) | 0.75 (0.08)
Statistical Analysis 1: Comparison: ChondroCelect vs Microfracture; Test for superiority; Test type: Superiority or Other; p = 0.003, ANCOVA; Adjusted for age, associated lesion(s) and location of lesion

2. Primary Outcome: Overall Histology Assessment on First Subscale of ICRS II Score
Description: Overall histology assessment of cartilage repair, first subscale of International Cartilage Repair Society II (ICRS II) score by two blinded independant histopathologists on a visual analogue scale (VAS 0-100mm) from worst (0) to best (100)
Time Frame: 12 months post-surgery
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: Points on a scale
Arm/Group | ChondroCelect | Microfracture
Number analyzed (Participants) | 51 | 58
Points on a scale | 55.11 (3.98) | 44.20 (3.74)
Statistical Analysis 1: Comparison: ChondroCelect vs Microfracture; Test for superiority; Test type: Superiority or Other; p = 0.010, ANCOVA; Adjusted for age, associated lesion(s) and location of lesion

3. Primary Outcome: Change From Baseline in Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) at 12-18 Months (Average)
Description: Overall Knee injury and Osteoarthritis Outcome score (average of 4 KOOS subdomains, Sports not included) at the average of 12-18 months (calculated by averaging change from baseline measurements at 12 and 18 months). Best score = 100; worst score = 0. The analysis was the average of the change from baseline at the 12 and 18 months timepoints.
Time Frame: Average change from baseline in Overall KOOS at 12-18 months post-surgery
Population: FAS (with LOCF for treatment failures)
Measure: Least Squares Mean (Standard Error); unit: points on a scale (0-100)
Arm/Group | ChondroCelect | Microfracture
Number analyzed (Participants) | 51 | 58
points on a scale (0-100)
  Change in oKOOS | 16.18 (2.42) | 14.37 (2.35)
  Baseline value | 56.30 (13.61) | 59.53 (14.95)
  Value at 12 months | 73.26 (14.66) | 73.10 (16.01)
  Value at 18 months | 74.73 (17.01) | 75.04 (14.50)
Statistical Analysis 1: Comparison: ChondroCelect vs Microfracture; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -9 % points; ANCOVA; Adjusted for baseline Overall KOOS score, age, associated lesion(s) and location of lesion; Mean Difference (Final Values) = 1.81, 95% CI [-3.28 to 6.90], Standard Error of Mean 2.4

4. Secondary Outcome: Change From Baseline in Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) at 36 Months
Description: Overall Knee injury and Osteoarthritis Outcome score (average of 4 KOOS subdomains: Activities of Daily Living, Quality of Life, Symptoms and Stiffness Pain; Sports not included) at 36 months (change from baseline). Best = 100; worst = 0.
Time Frame: Change from baseline in Overall KOOS at 36 months post-surgery
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | ChondroCelect | Microfracture
Number analyzed (Participants) | 51 | 58
Units on a scale
  Change in oKOOS | 21.25 (3.60) | 15.83 (3.48)
  Baseline value | 56.30 (1.91) | 59.46 (1.98)
  Value at 36 month | 78.46 (18.70) | 74.47 (18.60)

5. Secondary Outcome: Number of Treatment Failures at 36 Months
Description: Participants with failed treatment - defined as the number of patients who underwent a reintervention of the index lesion - at 36 months.
  The index lesion is the lesion that was initially treated in the study.
Time Frame: Continuous
Measure: Number; unit: Participants
Arm/Group | ChondroCelect | Microfracture
Number analyzed (Participants) | 51 | 58
Participants | 2 | 7

6. Secondary Outcome: Safety: Adverse Events
Description: Side effects are recorded as the number of patients with adverse events. These events are coded according to the Medical Dictionary for Regulatory Affairs (MedDRA terms).
Time Frame: continuous up to 60 months
Measure: Number; unit: participants
Arm/Group | ChondroCelect | Microfracture
Number analyzed (Participants) | 51 | 58
participants | 51 | 61

7. Post Hoc Outcome: Change From Baseline in Overall Knee Injury and Osteoarthritis Outcome Score (KOOS) at 60 Months
Description: Patient-administered instrument to assess the patients opinion about their knee and associated problems. It consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life QOL. The last week is taken into consideration when answering questions. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. The result can be plotted as an outcome profile.
Time Frame: 60 months
Population: FAS population with imputation for treatment failures by LOCF
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ChondroCelect | Microfracture
Number analyzed (Participants) | 43 | 55
units on a scale | 21.17 (2.89) | 14.07 (2.54)

8. Post Hoc Outcome: Number of Treatment Failures at 60 Months Post-surgery
Description: Participants with failed treatment - defined as the number of patients who underwent a reintervention of the index lesion - at 60 months.
  The index lesion is the lesion that was initially treated in the study.
Time Frame: 60 months
Measure: Number; unit: participants
Arm/Group | ChondroCelect | Microfracture
Number analyzed (Participants) | 51 | 58
participants | 7 | 10

ADVERSE EVENTS:
Time Frame: From baseline up to 36 months database lock
Description: The Intention To Treat population consists of 57 ChondroCelect patients and 61 microfracture patients.
  The FAS consists of 51 ChondroCelect and 61 microfracture patients. Since no events were reported for the 6 ChondroCelect randomized patients that were never treated, the results for the ChondroCelect group are presented for the FAS population.
Arm/Group | ChondroCelect | Microfracture
Serious Adverse Events (participants affected / at risk) | 10/51 | 12/61
Other Adverse Events (participants affected / at risk) | 50/51 | 51/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ChondroCelect (N=51) | Microfracture (N=61)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypersensitiviy (Immune system disorders) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myopia (Eye disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Testicular retraction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Anal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
perianal abscess (Infections and infestations) | 1 (1) | 0 (0)
hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
whiplash injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
arthralgia (knee pain) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ChondroCelect (N=51) | Microfracture (N=61)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 (38) | 37 (37)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 10 (10)
Bronchitis (Infections and infestations) | 6 (6) | 2 (2)
Cartilage hypertrophy (Musculoskeletal and connective tissue disorders) | 14 (14) | 8 (8)
Chondropathy (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Ear infection (Infections and infestations) | 3 (3) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 4 (4)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 3 (3)
Graft complication (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 11 (11)
Influenza (Infections and infestations) | 11 (11) | 16 (16)
Influenza-like illness (General disorders) | 5 (5) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 2 (2)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 10 (10) | 4 (4)
Joint effusion (Musculoskeletal and connective tissue disorders) | 13 (13) | 7 (7)
Joint sprain (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 11 (11) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Nasopharyngitis (Infections and infestations) | 14 (14) | 10 (10)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Pharyngitis (Infections and infestations) | 5 (5) | 5 (5)
Pyrexia (General disorders) | 5 (5) | 4 (4)
Sinusitis (Infections and infestations) | 4 (4) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Therapeutic product ineffective (General disorders) | 4 (4) | 9 (9)
Weight decreased (Investigations) | 3 (3) | 3 (3)
Weight increased (Investigations) | 3 (3) | 4 (4)
joint lock (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
cartilage injury (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less